CLINICAL TRIAL: NCT07204535
Title: Post-TRaUmatic STress Disorder Induced by Gynecological Brachytherapy
Acronym: TRUST-GB
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-004; 2025-A00672-47 (Other: ID-RCB number)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Brachytherapy; Post-TRaUmatic STress Disorder; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with cervical cancer with an indication for uterovaginal brachytherapy
  Interventions: Other: Prospective questionnaires

INTERVENTIONS:
Other: Prospective questionnaires — Post-traumatic stress disorder Checklist version DSM-5 (PCL-5) and quality of life questionnaires

SUMMARY:
This is a multicenter, prospective study aimed at providing information on the psychological effects (including post-traumatic stress symptoms) of utero-vaginal brachytherapy in patients with cervical cancer using self-administered questionnaires. The study also aims to assess the persistence of these symptoms over time, up to 5 years after brachytherapy. The results could help identify patients at risk of post-traumatic stress in this context and develop appropriate psychological interventions to improve their psychological well-being during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cervical cancer with an indication for High-dose rate (HDR) or pulse-dose rate (PDR) uterovaginal brachytherapy;
* Squamous cell carcinoma or other histological types;
* WHO ≤ 2;
* Ability to complete validated questionnaires in French;
* Informed consent to participate in the study;
* Patients over 18 years old

Exclusion Criteria:

* Inability to understand or respond to questionnaires due to a cognitive disorder, intellectual disability, language barrier, or psychiatric disorder that impairs judgment;
* Patient under juridic protection;
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patient with cervical cancer with an indication for High-dose rate (HDR) or pulse-dose rate (PDR) uterovaginal brachytherapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2030-10-27 (Estimated); Study Completion 2031-10-27 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder evaluation | at 2 months
  Evaluation with post-traumatic stress disorder Checklist version DSM-5 (PCL-5) - questionnaire with a Cut off score ≥ 32

SECONDARY OUTCOMES:
Anxiety and Depression | until 60 months
  Hospital Anxiety and Depression scale
Quality of Life (general module) | until 60 months
  Evaluated with EORTC QLQ-C30 questionnaire
Quality of Life (cervical cancer module) | until 60 months
  Evaluated with EORTC QLQ-CX24 questionnaire
Sexual Health evaluation | until 60 months
  Sexual Health Questionnaire (EORTC SHQ-22)

CONTACTS AND LOCATIONS:
Overall Officials: George NOEL, MD, PhD, Principal Investigator — ICANS, CPS
Locations (1):
- ICANS, Strasbourg, France